CLINICAL TRIAL: NCT01627873
Title: Effect of Remifentanil on Postoperative Cognitive Function in Patients Undergoing Major Abdominal Surgery
Brief Title: Effect of Remifentanil on Postoperative Cognition Function in Patients Undergoing Major Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Germano De Cosmo, Germano De Cosmo, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: A/575/2009
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Patients Undergoing Major Abdominal Surgery; Postoperative Confusion
Keywords: Major abdominal surgery; analgesic method; Fentanyl; Remifentanyl; Postoperative cognitive disorder; Pro and anti inflammatory cytokines
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Remifentanil; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanyl (Experimental): In group A induction of anesthesia will be performed with Propofol (2mg/kg), Cisatracurium (0.15mg/kg)and continous infusion of Remifentanil (0.15mcg/kg/min).Anesthesia will be maintained by Sevoflurane with oxygen (Fi=40%)and air, with a MAC value to maintain BIS between 40 and 60. Intraoperative analgesia will be obtained with Remifentanil 0.15-0.25mcg/kg/min. Additional boluses of Cisatracurium (0.02mcg/kg)will be administered as needed during surgery. At the beginning of closure of the peritoneum bolus of morphine (0.1mg/kg)and acetaminophen 1g will be administered. Propofol and remifentanil infusions will be interrupted at the end of wound closure.
  Interventions: Drug: Remifentanil
- Fentanyl (Active Comparator): In group B anesthesia will be induced by Propofol (2mg/kg), Fentanyl (2mcg/kg)and Cisatracurium (0.15mg/kg). Anesthesia will be maintained by Sevoflurane, oxygen (Fi=40%) and air and boluses of Fentanyl (50mcg). additional boluses of Cisatracurium (0.02mg/kg)will be administered as needed during surgery. At the beginning of closure of the peritoneum acetaminophen 1g will be administered.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — In group A induction of anesthesia will be performed with Propofol (2mg/kg), Cisatracurium (0.15mg/kg)and continous infusion of Remifentanil (0.15mcg/kg/min).Anesthesia will be maintained by Sevoflurane with oxygen (Fi=40%)and air, with a MAC value to maintain BIS between 40 and 60. Intraoperative analgesia will be obtained with Remifentanil 0.15-0.25mcg/kg/min. Additional boluses of Cisatracurium (0.02mcg/kg)will be administered as needed during surgery. At the beginning of closure of the peritoneum bolus of morphine (0.1mg/kg)and acetaminophen 1g will be administered. Propofol and remifentanil infusions will be interrupted at the end of wound closure.
  Arms: Remifentanyl
Drug: Fentanyl — In group B anesthesia will be induced by Propofol (2mg/kg), Fentanyl (2mcg/kg)and Cisatracurium (0.15mg/kg). Anesthesia will be maintained by Sevoflurane, oxygen (Fi=40%) and air and boluses of Fentanyl (50mcg). additional boluses of Cisatracurium (0.02mg/kg)will be administered as needed during surgery. At the beginning of closure of the peritoneum acetaminophen 1g will be administered.
  Arms: Fentanyl

SUMMARY:
The purpose of this study is to investigate the effects of two different analgesic methods (Fentanyl vs Remifentanil) during major abdominal surgery on postoperative cognitive status of patients.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of two different analgesic methods (Fentanyl vs Remifentanil) during major abdominal surgery on postoperative cognitive status of patients. In particular, whether there is a correlation between type of anesthesia and the appearance of postoperative cognitive disorder (POCD), including type of anesthesia and levels of pro and anti inflammatory cytokines and investigate whether there is an association between presence or absence of POCD and cytokines levels

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years
* Patients undergoing major abdominal surgery, in General Anesthesia
* ASA class status I-III

Exclusion Criteria:

* History of allergy to drugs used in the study
* Mini-Mental State Examination (MMSE) value < 26
* Expected duration of anesthesia less than 1 hour and more than 4 hours
* Presence of a cognitive disorder severity of overt such as to prevent collaboration of the patient
* Presence of severe electrolyte disturbances or not controlled bool glucose levels
* History of pain or cerebral vascular disease on the basis of significant carotid or cerebral artery stenosis, to be verified by scanning eco-color doppler
* Habitual use of tranquillizers or other drugs affecting the central nervous system
* Difficulties in the management of the airways, such as to make the necessary changes in anesthesia technique
* Severe hypotension or hypertension or other vascular disorders, particularly thrombotic events or bleeding during surgery or in the perioperative period
* Bleeding that requires blood transfusion
* Medication needs higher or lower than that indicated in the protocol to ensure the depth of hypnosis, indicated by values of BIS targets
* Refusal by the patient

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rey verbal memory test of words before and after major abdominal surgery | participants will be followed the day before and after surgery and for the duration of hospital stay, an expected average of 5 days
  In test of Rey to the subject is presented for 5 times the same list of 15 bisyllabic words or trisillabic common use of which he must recall as many as possible within 1 minute; after about 15 minutes the patient, meanwhile distracted by the test , must again try to remember the greatest number possible without a further reading. The maximum possible score of the first phase of the test is an expression of the ability of short term memory of the subject, the result of the test is repeated at a distance of 15 minutes is indicative of its storage capacity, to intermediate term.
Stroop Test before and after surgery | participants will be followed the day before and after surgery and for the duration of hospital stay, an expected average of 5 days
  In the Stroop Test patient is instructed to read a random sequence of adjectives "green", "red", "blue" written in black font, then he refers the colour of a succession of circumferences filled of the three colors above in random order; finally, another random succession of three words "green", "red", "blue" written in three characters of the same colors, but not associated with corresponding adjective. Number of errors that the subject does in reading is an indication of its ability to attention

SECONDARY OUTCOMES:
Quantitative determination of serum pro and anti inflammatory cytokines before and after surgery | participants will be followed the day before and after surgery and for the duration of hospital stay, an expected average of 5 days
  Blood samples will be made for the quantitative determination of serum cytokines IL-1β, IL-6, IL-8, TNF-α, IL-10 and IL-12. Determinations will be given by Multiplex Elisa method.

CONTACTS AND LOCATIONS:
Overall Officials: Germano De Cosmo, Associated Professor, Study Director — Catholic University of the Sacred Heart - Rome
Locations (1):
- Policlinico Universitario "A.Gemelli", Rome, Rome, Italy

REFERENCES:
- [Background] Rasmussen LS, Moller JT. Central nervous system dysfunction after anesthesia in the geriatric patient. Anesthesiol Clin North Am. 2000 Mar;18(1):59-70, vi. doi: 10.1016/s0889-8537(05)70149-8. PMID 10935000
- [Background] Dodds C, Allison J. Postoperative cognitive deficit in the elderly surgical patient. Br J Anaesth. 1998 Sep;81(3):449-62. doi: 10.1093/bja/81.3.449. No abstract available. PMID 9861139
- [Background] Rasmussen LS. Perioperative cognitive decline: the extent of the problem. Acta Anaesthesiol Belg. 1999;50(4):199-204. No abstract available. PMID 10603995
- [Background] Parikh SS, Chung F. Postoperative delirium in the elderly. Anesth Analg. 1995 Jun;80(6):1223-32. doi: 10.1097/00000539-199506000-00027. PMID 7762856
- [Background] Moller JT. Cerebral dysfunction after anaesthesia. Acta Anaesthesiol Scand Suppl. 1997;110:13-6. doi: 10.1111/j.1399-6576.1997.tb05484.x. No abstract available. PMID 9248516
- [Background] Diegeler A, Hirsch R, Schneider F, Schilling LO, Falk V, Rauch T, Mohr FW. Neuromonitoring and neurocognitive outcome in off-pump versus conventional coronary bypass operation. Ann Thorac Surg. 2000 Apr;69(4):1162-6. doi: 10.1016/s0003-4975(99)01574-x. PMID 10800812
- [Background] Wilson CJ, Finch CE, Cohen HJ. Cytokines and cognition--the case for a head-to-toe inflammatory paradigm. J Am Geriatr Soc. 2002 Dec;50(12):2041-56. doi: 10.1046/j.1532-5415.2002.50619.x. PMID 12473019
- [Background] Wan Y, Xu J, Ma D, Zeng Y, Cibelli M, Maze M. Postoperative impairment of cognitive function in rats: a possible role for cytokine-mediated inflammation in the hippocampus. Anesthesiology. 2007 Mar;106(3):436-43. doi: 10.1097/00000542-200703000-00007. PMID 17325501
- [Background] Buvanendran A, Kroin JS, Berger RA, Hallab NJ, Saha C, Negrescu C, Moric M, Caicedo MS, Tuman KJ. Upregulation of prostaglandin E2 and interleukins in the central nervous system and peripheral tissue during and after surgery in humans. Anesthesiology. 2006 Mar;104(3):403-10. doi: 10.1097/00000542-200603000-00005. PMID 16508385
- [Background] Winterhalter M, Brandl K, Rahe-Meyer N, Osthaus A, Hecker H, Hagl C, Adams HA, Piepenbrock S. Endocrine stress response and inflammatory activation during CABG surgery. A randomized trial comparing remifentanil infusion to intermittent fentanyl. Eur J Anaesthesiol. 2008 Apr;25(4):326-35. doi: 10.1017/S0265021507003043. Epub 2007 Nov 16. PMID 18005471
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Rohan D, Buggy DJ, Crowley S, Ling FK, Gallagher H, Regan C, Moriarty DC. Increased incidence of postoperative cognitive dysfunction 24 hr after minor surgery in the elderly. Can J Anaesth. 2005 Feb;52(2):137-42. doi: 10.1007/BF03027718. PMID 15684252
- [Background] Collie A, Darby DG, Falleti MG, Silbert BS, Maruff P. Determining the extent of cognitive change after coronary surgery: a review of statistical procedures. Ann Thorac Surg. 2002 Jun;73(6):2005-11. doi: 10.1016/s0003-4975(01)03375-6. PMID 12078822